CLINICAL TRIAL: NCT04066959
Title: Improving Diabetes Health in Emerging Adulthood Through an Autonomy Supportive Intervention
Brief Title: Improving Diabetes in Emerging Adulthood
Acronym: IDEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, April Carcone, Associate Professor, Wayne State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: R01DK116901 (NIH); 1R01DK116901-01A1 (NIH)
Record Dates: First submitted 2019-07-24; First posted 2019-08-26 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: emerging adults; ehealth intervention; diabetes; diabetes management; adolescents; self-determination theory
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The study will use an 8-arm full factorial design. In arms 1-3 participants will receive 1 of the 3 intervention components, arms 4-6 receive a combination of 2 components, arm 7 receives all 3 components, and arm 8 is the standard care control. The study will use the mixed effects linear model for the ANOVA of a factorial design powered on the main effects to identify the intervention components that significantly contribute to a clinically significant improvement in HbA1c. Each model will include a random intercept and slope and fixed effects for treatment combinations and time, as well as the stratification variable. The component selection experiment will result in empirical evidence supporting the efficacy of an autonomy support intervention composed of one or more components to improve metabolic control.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor/data collector will be kept blind to treatment assignments to the extent possible in a behavioral trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Question Prompt List (QPL) (Experimental): A QPL is a simple, inexpensive communication tool that is comprised of list of questions related to the physical and psychosocial aspects of an illness and treatment components about which patients may want to ask their diabetes care team during a routine diabetes clinic visit.
  Interventions: Behavioral: Question Prompt List (QPL)
- Motivation Enhancement System (MES) (Experimental): MES is a brief, 2-session computer-delivered intervention to enhance intrinsic motivation for behavior change. MES is grounded in the Motivational Interviewing framework and the Information-Motivation-Behavioral Skills model of health behavior change. Session 1 begins with psychoeducation describing optimal diabetes self-management, then youth motivation for diabetes self-management is assessed and followed by exercises designed to increase or reinforce his/her current motivational state (e.g., decisional balance) and build self-efficacy, (e.g., building on strengths and past success). Session 1 concludes with goal setting to promote autonomous diabetes self-management. Session 2 begins with an assessment of progress toward the behavioral goal and proceeds to build motivation and self-efficacy with exercises consistent with the youth's current motivational state. Session 2 concludes with goal setting to promote autonomous diabetes self-management.
  Interventions: Behavioral: Motivational Enhancement System (MES)
- Text Message Reminders (TXT) (Experimental): Participants will receive 30 days of one-way text messages targeting one of three key daily diabetes care behaviors: monitoring blood glucose, insulin administration, or carbohydrate counting. Participants will set a reminder schedule, i.e., frequency and timing of text message reminders.
  Interventions: Behavioral: Text Message Reminders (TXT)
- QPL & MES (Experimental): Participants will receive the QPL and MES interventions as described above.
  Interventions: Behavioral: Motivational Enhancement System (MES); Behavioral: Question Prompt List (QPL)
- QPL & TXT (Experimental): Participants will receive the QPL and TXT interventions as described above.
  Interventions: Behavioral: Question Prompt List (QPL); Behavioral: Text Message Reminders (TXT)
- MES & TXT (Experimental): Participants will receive the MES and TXT interventions as described above.
  Interventions: Behavioral: Motivational Enhancement System (MES)
- MES, QPL & TXT (Experimental): Participants will receive the MES, QPL, and TXT interventions as described above.
  Interventions: Behavioral: Motivational Enhancement System (MES); Behavioral: Question Prompt List (QPL); Behavioral: Text Message Reminders (TXT)
- Standard Medical Care (No Intervention): Participants will receive standard medical care at one of two participating clinical sites. Clinical practices at these sites are consistent with the standards of T1D care recommended by the American Diabetes Association and will include diabetes clinic visits every 3-4 months for routine diabetes medical care provided by an endocrinologist and/or nurse practitioner.

INTERVENTIONS:
Behavioral: Motivational Enhancement System (MES) — MES is a brief eHealth intervention delivered via an internet-based software application. MES is grounded in the Motivational Interviewing framework and the Information-Motivation-Behavioral Skills model of health behavior change. The goal of MES is to increase motivation to complete daily diabetes care tasks. MES consists of two 20-minute sessions that integrate psychoeducation with motivation-enhancing therapeutic exercises and behavioral goal setting.
  Arms: MES & TXT; MES, QPL & TXT; Motivation Enhancement System (MES); QPL & MES
Behavioral: Question Prompt List (QPL) — A QPL is a list of questions related to the physical and psychosocial aspects of diabetes and treatment that youth may want to ask their physicians during a clinic visit. The theoretical foundation for the QPL resides in social-cognitive theory which posits that behavioral performance is a function of self-efficacy and behavioral expectations. Thus, the goal of a QPL is to increase self-efficacy and active participation in clinical care. QPL is completed within 14-days of a diabetes clinic visit and results in a personalized set of questions for youth to bring to their clinic visit.
  Arms: MES, QPL & TXT; QPL & MES; QPL & TXT; Question Prompt List (QPL)
Behavioral: Text Message Reminders (TXT) — TXT is a behavioral support strategy composed of one-way text message reminders to promote daily diabetes care task completion. TXT is supported by social cognitive theory which suggests that consistent task completion leads to perceptions of control and supports goal attainment. TXT may also foster a stronger relationship with diabetes care providers through greater communication and satisfaction. Youth will receive daily reminders to complete key diabetes care tasks.
  Arms: MES, QPL & TXT; QPL & TXT; Text Message Reminders (TXT)

SUMMARY:
This project will test the efficacy of a multi-component behavioral intervention to improve metabolic control among older adolescents and emerging adults (16-21) with T1D, a group with chronic poor metabolic control. This intervention is grounded in self-determination theory which states that a youth who believes their diabetes management is self-directed, competent, and supported by others is more likely to consistently complete their diabetes self-care. This theory-driven intervention will be scalable to a variety of chronic illness contexts and the knowledge gained from this research will inform self-determination theory and different interventions targeting this population (currently there are no interventions that directly target emerging adults).

DETAILED DESCRIPTION:
This project will use the multiphase optimization strategy (MOST) approach to test the efficacy of an autonomy supportive behavioral intervention to improve metabolic control among older adolescents and emerging adults (16-25) with T1D. Youth this age demonstrate chronic poor metabolic control that persists into adulthood leading to the premature emergence of short- and long-term diabetes complications. Developmentally, adolescence and emerging adulthood is a time when the need for independence and autonomy are particularly salient. This new intervention will leverage youths' desire for autonomy by designing an intervention to support diabetes self-management autonomy. This intervention is guided by self-determination theory (SDT) which suggests that autonomous (i.e., self-initiated, driven by intrinsic versus extrinsic motivation) diabetes management depends upon three conditions: 1) the perception that one's behavior is self-directed, 2) feelings of competence, or self-efficacy, and 3) the existence of caring relationships supportive of the behavior. The investigators have identified three intervention components that target the SDT constructs. A question prompt list (QPL) is a simple, inexpensive tool comprised of a list of questions that patients might consider asking their health care provider during a clinic visit. QPLs empower patients to assume a more active role (asking questions and stating concerns) during clinic visits. The Motivation Enhancing System (MES) is an eHealth intervention to increase intrinsic motivation for health behavior change. MES content is based on the Motivational Interviewing (MI) framework and the Information-Motivation-Behavioral Skills (IMB) model of health behavior change which posits that behavior change results from the joint function of three critical components: accurate information about risk behaviors or their replacement health behaviors, motivation to change behavior, and behavioral skills necessary to perform the behavior (self-efficacy). Text message reminders (TXT) are a strategy to encourage youth to complete their diabetes self-care that also lead to gains in self-efficacy and a stronger relationship with diabetes care providers through greater communication and satisfaction. The investigators will test the efficacy of these intervention components toward improving metabolic control in a component selection experiment (N=320). The experiment will use a full factorial research design with random assignment to determine which intervention components contribute to a clinically significant improvement (≥0.5%) in HbA1c. The result of this research will be an optimized, multi-component intervention with effect size estimates that will be used to inform a large scale, fully powered effectiveness trial. This theory-driven intervention will be scalable to a variety of chronic illness contexts and the knowledge gained from this research will inform self-determination theory and behavioral interventions targeting this population (for which there currently are none).

ELIGIBILITY:
Inclusion:

1. Age 16 years, 0 months - 25 years, 11 months
2. Type 1 diabetes (T1D)
3. HbA1c ≥7.5% currently and averaged over the previous 6 months
4. Duration of diabetes ≥6 months
5. English fluency, both verbal and written
6. Cell phone access with texting capability

   Exclusion:
7. Psychosis (e.g., schizophrenia or bipolar disorder)
8. Suicidal
9. Developmental delay (moderate or severe mental retardation, or autism) or reading level below sixth grade
10. The presence of another physical health condition that results in atypical diabetes management (e.g., cystic fibrosis)

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 113 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | Change from Baseline at 3 months (end of treatment) and change from baseline at 6 months (post-treatment)
  Hb1Ac will be obtained by using the Accubase A1c test kit.

SECONDARY OUTCOMES:
Diabetes Management Scale | Change from Baseline at 3 months (end of treatment) and change from baseline at 6 months (post-treatment)
  The Diabetes Management Scale (DMS) is a self-report measure of daily diabetes care that assesses a broad range of management behaviors, including insulin management, dietary management, blood glucose monitoring, and symptom response with good internal consistency (α=.74 to .84). Each item asks "What percent of the time do you (take your insulin)?" The response scale is 0-100%. A total score is obtained by summing the items to reflect overall management behavior.
Blood glucose testing | Change from Baseline at 3 months (end of treatment) and change from baseline at 6 months (post-treatment)
  The mean daily frequency of blood glucose testing during the 14 days prior to assessment downloaded from blood glucose meters.

CONTACTS AND LOCATIONS:
Overall Officials: April Carcone, PhD, Principal Investigator — Wayne State University
Locations (1):
- Detroit Medical Center, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Idalski Carcone A, Ellis DA, Eggly S, MacDonell KE, Ghosh S, Buggs-Saxton C, Ondersma SJ. Improving Diabetes Management in Emerging Adulthood: An Intervention Development Study Using the Multiphase Optimization Strategy. JMIR Res Protoc. 2020 Oct 20;9(10):e20191. doi: 10.2196/20191. PMID 33079068
- See also: Principal Investigator-hosted website to share the dissemination products from the research. — https://ideaproject.med.wayne.edu/publications